CLINICAL TRIAL: NCT02453243
Title: Emergency Department Safety Assessment and Follow-up Evaluation 2
Acronym: ED-SAFE-2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Massachusetts, Worcester (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Edwin Boudreaux, Vice Chair, Director of Research, University of Massachusetts, Worcester
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: H000007010; R01MH106726 (NIH)
Record Dates: First submitted 2015-04-16; First posted 2015-05-25 (Estimated); Last update posted 2020-08-07 (Actual); Status verified 2020-08

CONDITIONS: Suicide
Keywords: Suicide screening in the ED; Safety Planning
MeSH Terms: conditions — Suicide

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Baseline (No Intervention): Retrospective Chart Reviews will be conducted for the period between the original ED-SAFE and the new study to test the long-term sustainability of nurse administered universal screening implemented in the original study.
- Intervention (Other): 1. Safety Plan Intervention: Clinician training in safety planning, and
  2. A Lean Implementation Strategy: The Implementation of the safety planning guided by Lean
  Combine, this is expected to increase safety planning by clinicians.
  Interventions: Behavioral: Safety Planning; Behavioral: A Lean Implementation Strategy
- Maintenance (No Intervention): Test sustainability of safety planning during the Maintenance phase.

INTERVENTIONS:
Behavioral: Safety Planning — Suicide screen-positive patients who are to be discharged from the ED will receive personalized safety planning by a mental health clinician or nurse
  Arms: Intervention
Behavioral: A Lean Implementation Strategy — The Safety Planning Intervention will be implemented using Lean performance improvement strategies.
  Sites will be trained on the Safety Planning Intervention and Lean.
  Arms: Intervention

SUMMARY:
Many patients at risk for suicide are discharged from the ED with little or no intervention. Evidence-based suicide prevention interventions, like universal screening and safety planning should be adopted in clinical practice to help prevent suicidal behavior. This study will test the long-term sustainability of the nurse administered universal screening implemented in the original ED-SAFE study. Also, the investigators will test the impact of a new personalized Safety Planning Intervention guided by Lean has on suicide composite outcomes.

The ED-SAFE-2 will use a stepped wedge design where the original eight ED-SAFE sites will collect quantitative and qualitative data during the three phases: Baseline, Implementation, and Maintenance. Using this data, the ED-SAFE-2 will examine both within and between site differences for existing screening practices and new care processes, including safety planning. Most of the data collection on outcomes will be done by retrospective chart review.

A Lean Implementation Strategy will be used to ensure that adoption of improved care processes are fully supported vertically and horizontally within the organization, infrastructure is built that supports the efforts, and that the protocols fit naturally within roles, responsibilities, and clinical flow.

Consistent with the RFA's emphasis, the intervention target will be the clinician's behavior, including, at minimum, screening and safety planning. All emergency mental health and nursing personnel at the sites will be trained on safety planning, and Lean will be used to help ensure the safety planning is being implemented properly and consistently. The mechanisms of action of the combination of the safety planning training and Lean will be studied, allowing the team to establish both the effect the intervention has on the intervention target but also on the mechanisms of action comprised of departmental culture change and infrastructure support.

DETAILED DESCRIPTION:
Suicide risk is much more prevalent among general emergency department (ED) patients than in the general community but this risk often goes undetected, especially among patients presenting with non-psychiatric complaints. By definition, universal screening is the only way to identify occult risk among patients presenting for non-psychiatric complaints. Until recently, however, little was known about how to implement universal screening in a clinical ED setting or whether doing so had any effect on detecting risk. The ED-SAFE has shown that it is feasible to implement universal screening and that the screening increases detection of suicide risk.

Simply identifying risk is not sufficient; efforts must be taken to mitigate risk and prevent suicidal behavior. However, many studies have shown that even those patients identified as having clinically significant risk are often discharged home without receiving any kind of active intervention during the ED visit, with many not even receiving a psychiatric evaluation.1-3 Brief interventions that are a good fit for the ED are needed. One such intervention has received strong research support and has already been accepted as a best practice in the United States Department of Veterans Affairs: Safety Planning Intervention.4 This intervention, however, has not been adopted in civilian EDs and little is known about how to effectively implement it, and whether doing so impacts suicide-related outcomes.

This study will address the following specific aims:

Aim 1: Test the long-term sustainability of nurse administered universal screening implemented in the original study across two new time periods. (a) The first is the period between the original ED-SAFE and the new study (ED-SAFE-2), which represents an ecologically valid "natural" state without any grant support, hereafter referred to as Baseline. (b) The second is the Maintenance phase of the new study, which will represent a time period spanning a minimum of four years after screening was initially implemented.

• Primary hypothesis: Sites that sustained high screening rates (intervention target) will sustain improved suicide risk detection (patient outcome) during each time period examined. Sustained screening practices will be mediated through ED organizational characteristics and enabling infrastructure (mechanisms of action).

Aim 2: Test the impact of implementing the new personalized Safety Planning Intervention for patients with suicide risk who are discharged from the ED.

• Primary hypotheses: Clinician training in safety planning, combined with implementation guided by Lean, is expected to increase safety planning by clinicians (intervention target), which will result in reduced suicide and suicide-related acute healthcare in the 6-months post-visit (suicide composite outcome). This will be more likely in sites with organizational characteristics and infrastructure that supports safety planning (mechanisms of action).

Aim 3: Test sustainability of safety planning during the Maintenance phase.

• Primary hypotheses: Sustained safety planning will result in sustained reductions in the suicide composite outcome. Sustained safety planning will be mediated by strong organizational characteristics and a robust enabling infrastructure supporting safety planning.

ELIGIBILITY:
Inclusion Criteria:

* ED patients >18 years old
* Seen in ED triage

Exclusion Criteria:

* patients <18 years old
* not seen in ED triage
* Adults unable to consent
* Prisoners

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14250 (Actual)
Dates: Start 2014-01 (Actual); Primary Completion 2018-10 (Actual); Study Completion 2018-10 (Actual)

PRIMARY OUTCOMES:
Suicide Risk Screening | up to 4 years
  Consistent with the parent ED-SAFE, a completed suicide screen will be defined as any chart documentation of the presence OR absence of suicidal ideation AND presence or absence of a past suicide attempt (0 = None documented, 1 = Partial (+/- ideation OR attempt noted), 2 = Complete (+/- ideation AND attempt noted). The proportion of general ED patients with a complete screen within each study phase will comprise the primary clinician-level outcome for analyses pertaining to screening (Aim 1). Sensitivity analyses will expand the definition to partial OR complete screens.
Suicide Risk Detection | up to 4 years
  Using the parent ED-SAFE criteria, a positive screen (i.e., detection) will be defined as any individual who either endorsed active ideation OR reported a lifetime suicide attempt. The proportion of general ED patients with a positive screen within each study phase will comprise the primary patient-level outcome for analyses pertaining to risk detection.
Safety Planning & Suicide Composite | 6 months after the Index ED Visit
  We decided that our primary outcome measure should be a broadly defined composite that reflects the subsequent occurrence of significant suicidal behavior/risk. This measure will be defined as the occurrence of any one of the following: (a) suicide, (b) any ED visit or hospitalization related to suicidal ideation or behavior.

CONTACTS AND LOCATIONS:
Overall Officials: Edwin D Boudreaux, PhD, Principal Investigator — University of Massachusetts, Worcester
Locations (8):
- United States (8):
  - Maricopa Medical Center, Phoenix, Arizona
  - University of Arkansas Medical Center, Little Rock, Arkansas
  - University of Colorado Hospital, Aurora, Colorado
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Marlborough Hospital, Marlborough, Massachusetts
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Ohio State Univeristy Medical Center, Columbus, Ohio
  - Memorial Hospital of Rhode Island, Pawtucket, Rhode Island

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Boudreaux ED, Larkin C, Vallejo Sefair A, Ma Y, Li YF, Ibrahim AF, Zeger W, Brown GK, Pelletier L, Miller I; ED-SAFE 2 Investigators. Effect of an Emergency Department Process Improvement Package on Suicide Prevention: The ED-SAFE 2 Cluster Randomized Clinical Trial. JAMA Psychiatry. 2023 Jul 1;80(7):665-674. doi: 10.1001/jamapsychiatry.2023.1304. PMID 37195676